CLINICAL TRIAL: NCT02930174
Title: EIT Assessment of Lung Volume and Tidal Distribution: A Comparison of Non-Invasive Ventilation Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Carl Haas, Education & Research Coordinator, Respiratory Care, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HUM00102144
Record Dates: First submitted 2015-08-24; First posted 2016-10-12 (Estimated); Results first posted 2019-04-22 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Spontaneous Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Respironics V-60, then Draeger V500 (Active Comparator): Testing by applying noninvasive positive pressure ventilation (NPPV) via two different bilevel positive airway pressure (BiPAP) devices . Arm one applies the Respironics V-60, then the Drager V-500.
  Interventions: Device: noninvasive positive pressure ventilation
- Draeger V500, then Respironics V-60 (Active Comparator): Testing by applying noninvasive positive pressure ventilation (NPPV) via two different bilevel positive airway pressure (BiPAP) devices . Arm two applies the Drager V-500, then the Respironics V-60.
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive positive pressure ventilation — Application of various levels of positive pressure

SUMMARY:
This study is being done to further the investigators' knowledge of the EIT system and to see if measures between two non-invasive ventilation systems routinely used clinically are equivalent.

DETAILED DESCRIPTION:
Mechanical ventilation is life-saving technology but it can also inadvertently induce lung injury and increase morbidity and mortality. There currently is not an easy method of assessing the impact ventilator settings have on the degree of lung inflation. Computed tomography (CT), the gold standard for visually monitoring lung function, can provide detailed regional information of the lung. Unfortunately, it necessitates moving critically ill patients to a special diagnostic room and involves exposure to radiation like an X-ray.

A technique introduced in the 1980's, electrical impedance tomography (EIT), can non-invasively provide similar monitoring of lung function, and without the exposure to radiation. This imaging technique applies small alternating currents of electricity to surface electrodes to construct cross-sectional images of the lung.

Over that past several decades EIT has moved from the research lab to commercially available devices that are used at the bedside. EIT has also been applied to study the effects of various devices used to provide non-invasive ventilation. EIT may prove useful to optimally adjust non-invasive ventilation settings to improve ventilation and oxygenation. One such EIT system is manufactured by Draeger Medical. It is available in Europe and Canada but is not yet FDA approved for use in the United States.

This study is being done with healthy volunteers to further the investigators' knowledge of the EIT system and to see if measures between two non-invasive ventilation systems routinely used clinically are equivalent.

As this is a preliminary study looking at the EIT system vs 2 other devices, outcomes measures may be modified as the study progresses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older

Exclusion Criteria:

* Use of a cardiac pacemaker, an implantable cardioverter-defibrillator (ICD) or any other active implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-03-27 (Actual); Study Completion 2018-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Haas, MLS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were solicited via word of mouth from the medical staff and the respiratory therapy staff at our university hospital. Enrollment occurred from February 1, 2018 through March 27, 2018.
Pre-assignment Details: All volunteers were screened for any contraindication to applying the electrical impedance tomography device (pacemaker, etc) before signing an informed consent document. No volunteer had such contraindications and all were successfully studied.
Groups:
- Device 1, Then Device 2: Testing by applying noninvasive positive pressure ventilation (NPPV) via two different bilevel positive airway pressure (BiPAP) devices: Respironics V-60 (Device 1) and Drager V-500 (Device 2) in a crossover study
  Device 1 is a continuous high flow, blower type of generator.
- Device 2, Then Device 1: Testing by applying noninvasive positive pressure ventilation (NPPV) via two different bilevel positive airway pressure (BiPAP) devices: Respironics V-60 (Device 1) and Drager V-500 (Device 2) in a crossover study
  Device 2 is a critical care ventilator that has a specific NPPV mode.
Period: Overall Study
Arm/Group | Device 1, Then Device 2 | Device 2, Then Device 1
Started | 12 | 8
Completed | 12 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Device 1, Then Device 2: Testing by applying noninvasive positive pressure ventilation via two different bilevel positive airway pressure (BiPAP) devices: Respironics V-60 (Device 1) and Drager V-500 (Device 2)
  Device 1 is a continuous high flow, blower type of generator.
- Device 2, Then Device 1: Testing by applying noninvasive positive pressure ventilation via two different bilevel positive airway pressure (BiPAP) devices: Respironics V-60 (Device 1) and Drager V-500 (Device 2).
  Device 2 is a critical care ventilator that has a specific NPPV mode.
- Total: Total of all reporting groups
Arm/Group | Device 1, Then Device 2 | Device 2, Then Device 1 | Total
Number analyzed (Participants) | 12 | 8 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (13.2) | 43.8 (14.4) | 42.6 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 8 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 8 | 20

OUTCOME MEASURES:

1. Primary Outcome: Global Tidal Variation (TID)
Description: TID is the distribution of ventilation for a breath averaged over a defined section, the entire lung. TID is analogous to the tidal volume. Baseline is defined to be 100% and other measures are in comparison to baseline (eg, a value of 102 represents a 2% increase from baseline).
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of baseline
Groups:
- Respironics V-60: This device is a continuous high flow, blower type of generator.
- Draeger V-500: This device is an ICU ventilator
Arm/Group | Respironics V-60 | Draeger V-500
Number analyzed (Participants) | 20 | 20
percentage of baseline
  Baseline (no pressure) | 100 (0) | 100 (0)
  Continuous Positive Airway Pressure (CPAP) 5 | 101.7 (16.4) | 109.1 (22.1)
  Pressure Support (PS) 5, CPAP 5 | 131.8 (39.5) | 118.1 (32.8)
  PS 5, CPAP 10 | 128.6 (47.0) | 126.4 (45.5)
Statistical Analysis 1: Comparison: Respironics V-60 vs Draeger V-500; Test type: Equivalence — Two devices were tested while measuring the differences in lung impedance under multiple pressure settings to determine whether the devices perform in an equivalent fashion. We looked at the mean differences between the 2 devices across the 4 pressure settings; p = 0.26, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

2. Secondary Outcome: Regional Tidal Variation: Dorsal
Description: Distribution of ventilation for a breath averaged over a defined section, the dorsal lung regions. Reflects the percent of tidal volume distributed to that area.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of global TID
Groups:
- Drager V-500: This device is an ICU ventilator.
Arm/Group | Respironics V-60 | Drager V-500
Number analyzed (Participants) | 20 | 20
percentage of global TID
  Baseline (no pressure) | 56.8 (14.0) | 56.9 (12.4)
  CPAP 5 | 59.0 (19.4) | 60.9 (18.4)
  PS 5, CPAP 5 | 69.1 (31.1) | 61.5 (22.0)
  PS 5, CPAP 10 | 71.3 (39.8) | 67.0 (32.9)
Statistical Analysis 1: Comparison: Respironics V-60 vs Drager V-500; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.342, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

3. Secondary Outcome: Regional Tidal Variation: Ventral
Description: Distribution of ventilation for a breath averaged over a defined section, the ventral lung regions. Reflects the percent of tidal volume distributed to that area.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: percentage of global TID
Arm/Group | Respironics V-60 | Drager V-500
Number analyzed (Participants) | 20 | 20
percentage of global TID
  Baseline (no pressure) | 43.2 (14.0) | 43.2 (12.5)
  CPAP 5 | 42.62 (12.8) | 48.2 (21.0)
  PS 5, CPAP 5 | 61.5 (22.0) | 56.7 (25.7)
  PS 5, CPAP 10 | 67.0 (32.9) | 59.5 (24.9)
Statistical Analysis 1: Comparison: Respironics V-60 vs Drager V-500; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.184, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

4. Secondary Outcome: Global Change in End-expiratory Lung Impedance (EELI)
Description: EELI is the impedance at the end of tidal variation, or end-expiration. EELI reflects the end-expiratory lung volume (EELV); thus an increase in EELI represents and increase in lung volume.
  The change in EELI that the electrical impedance tomography (EIT) device (Pulmovista, Drager) provides is the percent difference between the EELI of a given period and the EELI during a baseline or reference period. Positive or negative percent change suggests an increase or decrease in EELI and presumably EELV by a similar percentage. The baseline measurements used here were taken breathing air and no pressures applied, while the other measurements were taken with varying levels of pressure applied.
  By definition, baseline is assigned the value of 0%, by the EIT device. While it would be helpful to have the actual numbers for the baseline impedance values, this data was not provided by the EIT device.
Time Frame: 1 day
Population: Because one subject's EELI data did not record properly on device 2, that subject's data was excluded from analysis for both arms.
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Respironics V-60 | Drager V-500
Number analyzed (Participants) | 19 | 19
percentage change from baseline
  Baseline (no pressure) | 0.00 (0.00) | 0.00 (0.00)
  CPAP 5 | 45.9 (28.9) | 70.7 (68.9)
  PS 5, CPAP 5 | 53.3 (33.3) | 61.0 (53.7)
  PS 5, CPAP 10 | 135.2 (65.6) | 141.0 (101.3)
Statistical Analysis 1: Comparison: Respironics V-60 vs Drager V-500; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.283, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

5. Secondary Outcome: Regional Change in EELI: Dorsal
Description: as for outcome 4
Time Frame: 1 day
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Groups:
- Respironics V-60: This device is a continuous high flow, blower type of generator (Respironics V-60).
Arm/Group | Respironics V-60 | Drager V-500
Number analyzed (Participants) | 19 | 19
percentage change from baseline
  Baleline (no pressure) | 0.00 (0.00) | 0.00 (0.00)
  CPAP 5 | 14.9 (13.8) | 18.7 (31.2)
  PS 5, CPAP 5 | 17.5 (15.8) | 12.0 (26.3)
  PS 5, CPAP 10 | 44.9 (27.3) | 36.4 (43.8)
Statistical Analysis 1: Comparison: Respironics V-60 vs Drager V-500; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.204, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

6. Secondary Outcome: Regional Change in EELI: Ventral
Description: as for outcome 4
Time Frame: 1 day
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage change from baseline
Arm/Group | Respironics V-60 | Drager V-500
Number analyzed (Participants) | 19 | 19
percentage change from baseline
  Baseline (no pressure) | 0.00 (0.00) | 0.00 (0.00)
  CPAP 5 | 31.0 (19.1) | 52.0 (47.9)
  PS 5, CPAP 5 | 35.8 (21.9) | 49.0 (40.2)
  PS 5, CPAP 10 | 90.3 (43.2) | 104.5 (72.8)
Statistical Analysis 1: Comparison: Respironics V-60 vs Drager V-500; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.136, ANOVA; Mean Difference (Final Values) = 0.1, Standard Deviation 2

ADVERSE EVENTS:
Time Frame: During study period (~90-120 minutes)
Groups:
- Volunteer: Testing by applying noninvasive positive pressure ventilation via two different bilevel positive airway pressure (BiPAP) devices: Respironics V-60 and Drager V-500.
  Respironics V-60: Continuous high flow, blower type of generator.
  Drager V-500: Critical care ventilator that has a specific NPPV mode.
Arm/Group | Volunteer
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT02930174/Prot_SAP_000.pdf